CLINICAL TRIAL: NCT05918081
Title: The Relationship of Aerobic Capacity With Agility, Core Muscle Endurance and Peripheral Muscle Strength in Adolescent Basketball Players
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Selva Otsay, Principal Investigator, Bezmialem Vakif University
Other Study IDs: BezmialemVU-KFR-SO-01
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Sports Physical Therapy
Keywords: Basketball; Aerobic Capacity; Agility; Core Muscle Endurance; Peripheral Muscle Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent Basketball Players: Adolescent male basketball players registered in a local basketball academy will form the universe of the research.
  Interventions: Other: Multi-Stage 20 m Shuttle Run Test

INTERVENTIONS:
Other: Multi-Stage 20 m Shuttle Run Test — The aerobic capacities of the participants will be evaluated with the Multi-Stage 20 m Shuttle Run Test, their agility levels with the Pro Agility Test, their core muscle endurance with the McGill Trunk Extensor and Flexor Endurance test and their peripheral muscle strength with the MicroFET® 2" handheld dynamometer.
  Other Names: Pro Agility Test; McGill Trunk Extensor and Flexor Endurance test; MicroFET® 2" handheld dynamometer

SUMMARY:
The aim of this study is to investigate the relationship of aerobic capacity with agility, core muscle endurance and peripheral muscle strength in adolescent basketball players.

DETAILED DESCRIPTION:
A basketball player must have good physical condition to contribute to the team. In this physical condition, especially cardiorespiratory endurance (aerobic and anaerobic capacity), agility, muscle endurance and strength are important for basketball.

Revealing the interaction of aerobic capacity, which is critical for basketball, with other physical fitness components such as agility, core muscle endurance and peripheral muscle strength may shed light on the shaping of basketball players' exercise programs.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 10-19
* Male gender
* Interested in basketball sport for at least one year

Exclusion Criteria:

* Refusing to participate in the study
* Having any disability (orthopedic, cardiovascular, etc.) that would prevent participation in the study

Ages: 10 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Adolescent Male Basketball Players
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity | One Month
  Maximum oxygen consumption (VO2max)

SECONDARY OUTCOMES:
Agility | One Month
  Time to complete the pro agility test
Core Muscle Endurance | One Month
  Mcgill trunk extensor and flexor muscle endurance test
Peripheral Muscle Strength | One Month
  Peripheral muscle strength to be evaluated with the MicroFET® 2" hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Selva Otsay, BPT, Principal Investigator — Bezmialem Vakif University; Semiramis Özyılmaz, PhD, Study Director — Bezmialem Vakif University; Gökhan C Törpü, BPT, Study Chair — Bezmialem Vakif University
Locations (1):
- Eyüp Basket Akademi, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mancha-Triguero D, Garcia-Rubio J, Antunez A, Ibanez SJ. Physical and Physiological Profiles of Aerobic and Anaerobic Capacities in Young Basketball Players. Int J Environ Res Public Health. 2020 Feb 21;17(4):1409. doi: 10.3390/ijerph17041409. PMID 32098230
- [Result] McInnes SE, Carlson JS, Jones CJ, McKenna MJ. The physiological load imposed on basketball players during competition. J Sports Sci. 1995 Oct;13(5):387-97. doi: 10.1080/02640419508732254. PMID 8558625